CLINICAL TRIAL: NCT02655263
Title: Substrate Metabolism, Growth Hormone Signaling (GH), and Insulin Sensitivity During GH and Ketone Bodies Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Ketone8000
Record Dates: First submitted 2016-01-07; First posted 2016-01-14 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — Human Growth Hormone; Ketone Bodies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): 12 hours of fasting
- GH infusion (Experimental): 12 hours of fasting
  Interventions: Drug: Somatropin
- GH and ketone bodies infusion (Experimental): 12 hours of fasting
  Interventions: Drug: Somatropin; Other: Ketone bodies

INTERVENTIONS:
Drug: Somatropin — Somatropin infusion (Genotropin®)
  Arms: GH and ketone bodies infusion; GH infusion
Other: Ketone bodies — ketone bodies infusion
  Arms: GH and ketone bodies infusion

SUMMARY:
Background: Humans naturally produce ketone bodies under daily living conditions. The main ketone bodies are two functioning acids, beta-hydroxybutyric acid (3-OHB) and acetoacetate, and the pH-neutral, but odorous, acetone. In the fed state, level of 3-OHB is suppressed to an almost unmeasurable level while, in the fasted state, it rises to 0.1-0.5 millimoles (mM). Main regulation of ketone synthesis is the abundance of sugars and resulting adaptations in insulin secretion. Thus, ketone bodies are formed when sugar is not readily available and insulin is suppressed. This picture is, to a certain degree, seen in acute inflammatory states and, indeed, during starvation, where level of 3-OHB increases to 5-8 mM.

Hypothesis:

1. Ketone bodies changes the insulin sensitivity and substrate metabolism in human subjects
2. Ketone bodies changes the GH signaling in muscle and adipose tissue

Aim: The investigators wish to provide knowledge on changes in metabolites and shift in signaling pathways and insulin sensitivity during GH infusion and concomitant ketone bodies infusion among healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* written consent
* body mass index (BMI) 18.5 - 25
* age 20-50 years

Exclusion Criteria:

* any kind of disease
* regular medication

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Insulin and growth hormone signaling, expressed as CHANGE in phosphorylation of intracellular target proteins in muscle- and fat-tissue. | Muscle and fat biopsies obtained at t1= 9.00 am (60 min) and t2=12.30 am (270 min) on each study day after 0, 4 and 8 weeks (interval of 4 weeks between each of the three study days
  Change in phosphorylation of target proteins using Western Blotting (WB)

SECONDARY OUTCOMES:
Glucose metabolism | Change in glucose metabolism using glucose tracer from t=0 min - 360 min on each study day after 0, 4 and 8 weeks (interval of 4 weeks between each of the three study days.
  Change in glucose metabolism assessed by tracer kinetics on every study day.
Insulin and growth hormone signaling, expressed as CHANGE in messenger ribonucleic acid (mRNA) expression of target genes in muscle- and fat-tissue. | Muscle and fat biopsies obtained at t1= 9.00 am (60 min) and t2=12.30 am (270 min) on each study day after 0, 4 and 8 weeks (interval of 4 weeks between each of the three study days.
  Change in mRNA expression of target genes using Polymerase Chain Reaction (PCR).
Investigation of the balance in the autonomic nervous system | Measurement of heart rate variability at t1=10.30 am(150 min) and 12.30 am (270 min) on each study day after 0, 4 and 8 weeks (interval of 4 weeks between each of the three study days.
  Heart rate variability (the study of beat-to-beat fluctuations in heart rate).

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L. Jørgensen, Professor, Principal Investigator — Aarhus University / Aarhus University Hospital; Jens Otto L. Jørgensen, Professor, Study Director — Aarhus University / Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Hogild ML, Hjelholt AJ, Hansen J, Pedersen SB, Moller N, Wojtaszewski JFP, Johannsen M, Jessen N, Jorgensen JOL. Ketone Body Infusion Abrogates Growth Hormone-Induced Lipolysis and Insulin Resistance. J Clin Endocrinol Metab. 2023 Feb 15;108(3):653-664. doi: 10.1210/clinem/dgac595. PMID 36240323